CLINICAL TRIAL: NCT03009396
Title: An Open Label Study to Assess the Efficacy and Safety of Fixed-Dose Combination RHB-104 in Subjects With Active Crohn's Disease Despite 26 Weeks of Participation in the MAP US RHB-104-01 Study
Brief Title: Open Label Efficacy and Safety of Anti-MAP (Mycobacterium Avium Ssp. Paratuberculosis) Therapy in Adult Crohn's Disease
Acronym: MAPUS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHB-104-04
Record Dates: First submitted 2016-12-26; First posted 2017-01-04 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease,; moderate to severe; remission; Mycobacterium avium paratuberculosis; antibiotic
MeSH Terms: conditions — Crohn Disease | interventions — Clarithromycin; Rifabutin; Clofazimine

STUDY DESIGN:
Intervention Model Description: Active
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RHB-104 - patients on ACTIVE therapy in RHB-104-01 study (Experimental): Subjects who were on the active therapy arm in the RHB-104-01 clinical study will continue to receive RHB-104 at 5 capsules twice a day in addition to the standard of care they received in the RHB-104-01 clinical study
  Interventions: Drug: RHB-104 (fixed-dose combination: 95 mg clarithromycin, 45 mg rifabutin, and 10 mg clofazimine)
- RHB-104 - patients on PLACEBO therapy in RHB-104-01 study (Experimental): Subjects who were on the active therapy arm in the RHB-104-01 clinical study will receive RHB-104 at 5 capsules twice a day in addition to the standard of care they received in the RHB-104-01 clinical study. The RHB-104 will be ramped up beginning at 1 capsule twice per day in week 1 increasing to 2 capsules twice per day in week 2, 3 capsules twice per day in week 3, 4 capsules per day in week 4 and achieving 5 capsules per day for the remainder of the study.
  Interventions: Drug: RHB-104 (fixed-dose combination: 95 mg clarithromycin, 45 mg rifabutin, and 10 mg clofazimine)

INTERVENTIONS:
Drug: RHB-104 (fixed-dose combination: 95 mg clarithromycin, 45 mg rifabutin, and 10 mg clofazimine) — For patients on ACTIVE or PLACEBO in the parent study (RHB-104-01), who were not in remission after 26 weeks
  Other Names: RHB-104

SUMMARY:
An open label extension to the RHB-104-01 Study.

DETAILED DESCRIPTION:
An Open Label Phase III Study to Assess the Efficacy and Safety of Fixed-Dose Combination RHB-104 in Subjects with Active Crohn's Disease Despite 26 Weeks of Participation in the MAP US RHB-104-01 Study.

ELIGIBILITY:
Inclusion Criteria:

* Signed fully informed consent (ICF) provided as per this protocol.
* Participation in RHB-104-01 for 26 weeks, and a Crohn's Disease Activity Index (CDAI) score of ≥ 150 at Visit Week 26.

OR

* More than 26 weeks, with a CDAI ≥150 at Visit Week 26 and all subsequent visits, and subject is between Week 26 and 52 within 4 weeks (28 days) of site activation (e.g. Subject with CDAI = 249 at week 26 and who is at week 38 at the time of site's activation for RHB-104-04 has a 4-week window to be enrolled in the open label study via the Optional Screening Visit)
* Current treatment with at least one of the following therapies which may be discontinued by the investigator as clinically indicated after 8 weeks of open label RHB-104 treatment:

  * Oral 5-acetyl salicylic acid (5-ASA) compounds
  * Azathioprine or 6-mercaptopurine (6-MP) or methotrexate
  * Infliximab or adalimumab OR Current treatment with corticosteroid therapy which must begin tapering after 4 weeks of treatment with open label RHB-104 (Refer to Appendix 13)
* White blood cell count ≥ 3.5x109 at screening (RHB-104-01 Visit Week 26 visit or Optional Screening visit)
* Subject agrees to use the following effective contraceptive methods

  * diaphragm, cervical cap, contraceptive sponge or condom) with spermicidal foam/gel/cream/suppository
  * IUD (intrauterine device) /IUS (intrauterine system)
  * progestogen injection (Depo-Provera®) throughout the study and for at least 6 weeks after last study drug administration, unless subject or partner of subject is post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation, or has had a vasectomy. Post-menopausal is defined as having experienced 12 consecutive months without menstruation.

In regions where local regulatory contraceptive requirements differ, the ICF (Informed Consent Form) will reflect local policies.

Exclusion Criteria:

1. Positive stool results for C. difficile.
2. Currently diagnosed or history of uveitis confirmed by either an ophthalmologist or optometrist.
3. Treatment with any medication that causes QT prolongation or Torsades de Pointes, including but not limited to: amiodarone, amitriptyline, astemizole, cisapride, citalopram dose greater than 20 mg/day, dihydroergotamine, disopyramide, dofetilide, dronedarone, ergotamine, ibutilide, ondansetron or other 5-HT3 (5-hydroxytryptamine three) receptor antagonists, pimozide, procainamide, quinidine, quinine, quinolones, ranolazine, risperidone, sotalol, terfenadine and tolterodine. QT prolonging drugs may be referenced at the CredibleMeds® web site: https://crediblemeds.org/index.php/drugsearch/
4. Treatment with the following CYP3A4 interactive medications: alfentanyl, alprazolam, amlodipine, anti-retroviral agents, apixaban, aprepitant, aripiprazole, atorvastatin, boceprevir, buspirone, carbamazepine, carvedilol, colchicine, cyclosporine, digoxin, diltiazem, estrogens, felodipine, fluconazole, fluvoxamine, grapefruit juice, haloperidol, ketoconazole, lovastatin, lurasidone, metoprolol, nefazodone, nifedipine, nisoldipine, nitrendipine, propranol, roflumilast, simvastatin, St. John's wort, and voriconazole.
5. Any evidence of any newly diagnosed significant hematological, hepatic, renal, cardiac, pulmonary, metabolic, neurological, psychiatric or other disease (e.g. porphyria) that might interfere with subject's ability to safely enter and or complete the study requirements.
6. Females who have a positive pregnancy test or are lactating.
7. Refusal to sign the study informed consent form.
8. Inability to be able to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study.
9. Clinically significant abnormalities of hematology or biochemistry as confirmed by repeat testing based on investigator's discretion, including but not limited to, elevations greater than 2 times the upper limit of normal of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) or creatinine clearance less than 60 ml/min at screening via estimated Cockcroft-Gault formula:

   Creatinine Clearance = [140 - age in years] * weight (kg) / 72 * Serum Creatinine (mg/dl) [multiply estimated rate by 0.85 for women], using actual body weight.
10. QTcF (shortening of the QT interval in the heart rate) >450ms in males and QTcF>460ms in females, bundle branch block, or major ST or T wave abnormalities that make the assessment of the QT impossible.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira N Kalfus, MD, Study Director — RedHill Biopharma Limited; David Y Graham, MD, Principal Investigator — Department of Medicine / Gastroenterology, Baylor College of Medicine, Houston
Locations (24):
- United States (6):
  - Digestive Care Associates, Inc., 1000 Laurel Street, San Carlos, California
  - Gastrointestinal Specialists of Georgia PC 711 Canton Rd. #300, Marietta, Georgia
  - Cotton-O'Neil Clinical Research Center, 720 SW Lane St., Topeka, Kansas
  - Chevy Chase Clinical Research, 5550 Friendship Blvd., Chevy Chase, Maryland
  - Commonwealth Clinical Studies, 189 Quincy St., Brockton, Massachusetts
  - ClinSearch 6035 Shallowford Road Suite 109, Chattanooga, Tennessee
- Discovery Clinical Services Ltd., 601 A Discovery St., Victoria, British Columbia, Canada
- Czechia (2):
  - Gastroenterologie s.r.o. Manesova 646, Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradecka poliklinika III Trida Edvarda Benese 1549/34, Hradec Králové
- Israel (3):
  - Ha'Emek Medical Center, Institute of Gastroenterology and Liver diseases, 21 Yitshak Rabin Boulevard, Afula
  - Gastroenterology Institute, Division of Medicine, Hadassah - Hebrew University Medical Center POB 12000, Jerusalem
  - Meir Medial Center, 59 Tchemacovsky St., Kfar Saba
- New Zealand (2):
  - Christchurch Hospital, 2 Riccarton Rd., Christchurch, Canterbury
  - Waikato Hospital, Department of Gastroenterology, Level B1, Menzies Building, Pembroke Street, Hamilton, Waikato Region
- Poland (7):
  - NZOZ Specjalistyczne Centrum Gastrologii GASTROMED, Wiejska 81, Bialystok
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej MSW W Gdańsku Oddział Gastroenterologiczny, Ul. Kartuska 4/6, Gdansk
  - UNICARDIA Specjalistyczne Centrum Leczenia Chorob Serca i Naczyn & UNIMEDICA. Specjalistyczne Centrum Medyczne Sp. z o.o., Kluczborska 15, Krakow
  - Wojewodzki Szpital Kliniczny w Olsztynie Oddzial Gastroenterologiczny, Zolnierska 18, Olsztyn
  - EuroMedis sp. z.o.o., Al. Powstancow Wielkopolskich 33a, Szczecin
  - Centralny Szpital Kliniczny MSW w Warszawie. Klinika Chorob Wewnetrznych i Gastroenterologii, Woloska 137,, Warsaw
  - ARS MEDICA s.c., Powstancow Slaskich 56A/2, Wroclaw
- Serbia (3):
  - Clinical Department of Gastroenterology and Hepatology Clinic for Internal Diseases Clinical Hospital Center Zvezdara Dimitrija Tucovica 161, Belgrade
  - Department of Gastroenterology and Hepatology, Clinical Hospital Center Zemun, Vukova 9, Belgrade
  - Center for Gastroenterohepatology, Clinic for Internal Medicine, Clinical Center Kragujevac, Zmaj Jovina 30, Kragujevac

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: RedHill home page — http://www.redhillbio.com

RESULTS

PARTICIPANT FLOW:
Groups:
- RHB-104 From RHB-104: RHB-104 (fixed-dose combination 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine): For patients who were in the RHB-104 arm but are not in remission after 26 weeks in the RHB-104-01 study.
- RHB-104 From Placebo: RHB-104 (fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine): For patients who were in the placebo arm but are not in remission after 26 weeks in the RHB-104-01 study.
Period: Overall Study
Arm/Group | RHB-104 From RHB-104 | RHB-104 From Placebo
Started | 16 | 38
Completed | 9 | 21
Not Completed | 7 | 17

BASELINE CHARACTERISTICS:
Population: Total Study
Groups:
- RHB-104: RHB-104; a fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine.
Arm/Group | RHB-104
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] — Age measured in years at Baseline Population: 16 subjects who transferred to the RHB-104-04 study were on RHB-104 in the RHB-104-01 (parent) study while 38 subjects were on placebo.
  years
    RHB-104 from RHB-104: number analyzed (Participants) | 16
    RHB-104 from RHB-104 | 48.6 (9.92)
    RHB-104 from placebo: number analyzed (Participants) | 38
    RHB-104 from placebo | 40.0 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 16 subjects who transferred to the RHB-104-04 study were on RHB-104 in the RHB-104-01 (parent) study while 38 subjects were on placebo.
  Participants
    RHB-104 from RHB-104: number analyzed (Participants) | 16
    RHB-104 from RHB-104: Female | 6
    RHB-104 from RHB-104: Male | 10
    RHB-104 from placebo: number analyzed (Participants) | 38
    RHB-104 from placebo: Female | 18
    RHB-104 from placebo: Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 16 subjects who transferred to the RHB-104-04 study were on RHB-104 in the RHB-104-01 (parent) study while 38 subjects were on placebo.
  Participants
    RHB-104 from RHB-104: number analyzed (Participants) | 16
    RHB-104 from RHB-104: American Indian or Alaska Native | 0
    RHB-104 from RHB-104: Asian | 0
    RHB-104 from RHB-104: Native Hawaiian or Other Pacific Islander | 0
    RHB-104 from RHB-104: Black or African American | 1
    RHB-104 from RHB-104: White | 15
    RHB-104 from RHB-104: More than one race | 0
    RHB-104 from RHB-104: Unknown or Not Reported | 0
    RHB-104 from placebo: number analyzed (Participants) | 38
    RHB-104 from placebo: American Indian or Alaska Native | 1
    RHB-104 from placebo: Asian | 0
    RHB-104 from placebo: Native Hawaiian or Other Pacific Islander | 0
    RHB-104 from placebo: Black or African American | 1
    RHB-104 from placebo: White | 36
    RHB-104 from placebo: More than one race | 0
    RHB-104 from placebo: Unknown or Not Reported | 0
Baseline Crohn's Disease Activity Index (CDAI) score [Mean (Standard Deviation); unit: units on a scale] — Generally, CDAI score can range from 0-approx. 600. (in this protocol up to 450) CDAI scores of 150-219 describe mildly active disease, while scores of 220-450 describe moderately active disease and score above 450 describe severe disease. Population: 16 subjects who transferred to the RHB-104-04 study were on RHB-104 in the RHB-104-01 (parent) study while 38 subjects were on placebo.
  units on a scale
    RHB-104 from RHB-104: number analyzed (Participants) | 16
    RHB-104 from RHB-104 | 295.42 (82.865)
    RHB-104 from placebo: number analyzed (Participants) | 38
    RHB-104 from placebo | 271.67 (58.379)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Remission at Week 16
Description: The number of patients who achieved a reduction of the total Crohn's Disease Activity Index (CDAI) score to less than 150 points.
  Lower CDAI scores indicate a better outcome.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Groups:
- RHB-104 From ACTIVE Arm of RHB-104-01: RHB-104; a fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine: For patients who were in the RHB-104 arm, but were not in remission after 26 weeks in the RHB-104-01 study.
- RHB-104 From PLACEBO Arm of RHB-104-01: RHB-104; a fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine: For patients who were in the placebo arm, but were not in remission after 26 weeks in the RHB-104-01 study.
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 16 | 38
Participants | 3 | 14

2. Secondary Outcome: Response at Week 16
Description: Reduction of the total Crohn's Disease Activity Index (CDAI) score by a minimum of 100 points Lower CDAI scores indicate a better outcome.
Time Frame: Week 16
Population: Number of subjects achieved response
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 16 | 38
Participants | 4 | 14

3. Secondary Outcome: The Number of Weeks for Patients to Achieve Remission
Description: [Date of first observed remission (CDAI less than 150) - date of first dose, or date of randomization if not dosed, plus 1] / 7 days. Subject who never experience remission during the study are censored at the time of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Number of subjects achieved remission, n (%) RHB-104 from RHB-104: 6 (37.5); RHB-104 from Placebo: 20 (52.6).
  Number of patients censored due to never achieving remission, n (%) RHB-104 from RHB-104: 10 (62.5); RHB-104 from Placebo: 18 (47.4)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 16 | 38
weeks | NA [NA to NA] — The value is not estimable. A 95% CI limit cannot be estimated based on Kaplan Meier methods used. | 25.1 [16.00 to 56.00]
Statistical Analysis 1: Comparison: RHB-104 From ACTIVE Arm of RHB-104-01 vs RHB-104 From PLACEBO Arm of RHB-104-01; Test type: Superiority; p = 0.2112, Log Rank

4. Secondary Outcome: Number of Weeks the Patients Are in Remission
Description: Duration of remission is defined as the number of weeks the subject is in remission (CDAI score < 150). It is calculated as the first date following remission at which CDAI is ≥150 minus the date of first remission, plus 1 day, divided by 7. Subjects who experienced remission and continued to be in remission at the time of their last CDAI assessment are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Reached duration of remission (dropped out of remission during the study), n (%): RHB-104 from RHB-104 5 (83.3); RHB-104 from Placebo: 8 (40.0). Number of patients censored due to remaining in remission during the study, n (%): RHB-104 from RHB-104 1 (16.7); RHB-104 from Placebo: 12 (60.0)
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- RHB-104 From PLACEBO Arm of RHB-104-01: RHB-104; a fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine: For patients who were in the placebo arm but are not in remission after 26 weeks in the RHB-104-01 study.
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 6 | 20
weeks | 11.7 [NA to NA] — The value is not estimable. A 95% CI limit cannot be estimated based on Kaplan Meier methods used | 45.0 [23.00 to NA] — The value is not estimable. A 95% CI limit cannot be estimated based on Kaplan Meier methods used.
Statistical Analysis 1: Comparison: RHB-104 From ACTIVE Arm of RHB-104-01 vs RHB-104 From PLACEBO Arm of RHB-104-01; Test type: Superiority; p = 0.0356, Log Rank

5. Secondary Outcome: Number of Weeks to Achieve Response
Description: [Date of first observed response (a reduction from baseline of ≥ 100 in CDAI score) - Date of first dose or date of randomization if not dosed + 1] / 7 Days. Subjects who never experienced response during the study are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Number of subjects achieved response, n (%): RHB-104 from RHB-104 5 (31.3); RHB-104 from Placebo 21 (55.3). Number of patients censored due to never achieving response, n (%): RHB-104 from RHB-104 11 (68.8); RHB-104 from Placebo 17 (44.7)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 16 | 38
Weeks | NA [16.14 to NA] — The value is not estimable. A 95% CI limit cannot be estimated based on Kaplan Meier methods used. | 26.1 [9.14 to 56.00]
Statistical Analysis 1: Comparison: RHB-104 From ACTIVE Arm of RHB-104-01 vs RHB-104 From PLACEBO Arm of RHB-104-01; Test type: Superiority; p = 0.0514, Log Rank

6. Secondary Outcome: Number of Weeks the Patients Are in Response.
Description: Duration of response is defined as the number of weeks the subject is in a state of response (a reduction from baseline of ≥ 100 in CDAI score). It is calculated as the first date following response at which the reduction from baseline in CDAI is <100 minus the date of first response, plus 1 day, divided by 7. Subjects who experienced response and continued to be in response at the time of their last CDAI assessment are censored at the date of their last CDAI assessment.
Time Frame: Baseline through week 52
Population: Reached duration of response (dropped out of response during the study), n (%): RHB-104 from RHB-104 3 (60.0); RHB-104 from placebo 7 (33.3). Number of patients censored due to remaining in response during the study, n (%): RHB-104 from RHB-104 2 (40.0); RHB-104 from placebo 14 (66.7)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 5 | 21
Weeks | 29.4 [10.86 to NA] — The value is not estimable. A 95% CI limit cannot be estimated based on Kaplan Meier methods used. | 45.0 [26.14 to NA] — The value is not estimable. A 95% CI limit cannot be estimated based on Kaplan Meier methods used.
Statistical Analysis 1: Comparison: RHB-104 From ACTIVE Arm of RHB-104-01 vs RHB-104 From PLACEBO Arm of RHB-104-01; Test type: Superiority; p = 0.1259, Log Rank

7. Secondary Outcome: Durable Remission Week 16 Through Week 52
Description: When a subject is in remission with a maximum CDAI score of 149 at every visit from week 16 through and including week 52.
Time Frame: Week 16 through week 52
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 16 | 38
Participants | 1 | 7
Statistical Analysis 1: Comparison: RHB-104 From ACTIVE Arm of RHB-104-01 vs RHB-104 From PLACEBO Arm of RHB-104-01; Test type: Superiority; p = 0.4114, Fisher Exact

8. Other Pre Specified Outcome: Increase in Milliseconds (ms) QT Wave
Description: The increase in the number of milliseconds change-from-baseline to week 52 in QTcF (Fridericia's Correction Formula of QT wave interval) (based on cardiac safety report).
Time Frame: week 52
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | RHB-104 From ACTIVE Arm of RHB-104-01 | RHB-104 From PLACEBO Arm of RHB-104-01
Number analyzed (Participants) | 8 | 18
ms | 23.9 [17.77 to 30.02] | 27.6 [23.66 to 31.63]

ADVERSE EVENTS:
Time Frame: Baseline through 30 days after last dose of study drug, or up to 13 months.
Groups:
- RHB-104 From RHB-104: RHB-104; a fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine: For patients who were in the RHB-104 arm but are not in remission after 26 weeks in the RHB-104-01 study.
- RHB-104 From Placebo: RHB-104; a fixed-dose combination of 95 mg clarithromycin, 45 mg rifabutin, 10 mg clofazimine: For patients who were in the placebo arm but are not in remission after 26 weeks in the RHB-104-01 study.
Arm/Group | RHB-104 From RHB-104 | RHB-104 From Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/16 | 4/38
Other Adverse Events (participants affected / at risk) | 14/16 | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHB-104 From RHB-104 (N=16) | RHB-104 From Placebo (N=38)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHB-104 From RHB-104 (N=16) | RHB-104 From Placebo (N=38)
Crohn's Disease (Gastrointestinal disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dental caries (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gingival discolouration (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Siliva discolouration (Gastrointestinal disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 2 | 9
Pollakiuria (Renal and urinary disorders) | 1 | 1
Weight decreased (Investigations) | 2 | 1
Weight increased (Investigations) | 2 | 1
Electrocardiogram abnormal (Investigations) | 1 | 1
Blood creatine phosphokinase abnormal (Investigations) | 1 | 0
Transaminases (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Inflective scleritis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Fatigue (General disorders) | 1 | 3
Pirexia (General disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03009396/SAP_000.pdf
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT03009396/Prot_001.pdf